CLINICAL TRIAL: NCT01049438
Title: A Prospective Trial of Nasal Mupirocin, Hexachlorophene Body Wash, and Systemic Antibiotics for Prevention of Recurrent Methicillin Resistant Staphylococcus Aureus Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Natividad Medical Center (Other)
Responsible Party: Allen Radner, MD, Navidad Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20020519
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Methicillin Resistant Staphylococcus Aureus Skin Infections
Keywords: MRSA; Methicillin Resistant Staphylococcus aureus; Staphylococcus aureus; Skin Infections; Body Decolonization
MeSH Terms: conditions — Staphylococcal Infections; Cellulitis | interventions — Triclosan; Trimethoprim, Sulfamethoxazole Drug Combination; Doxycycline; Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nasal, body, and systemic decolonization (Experimental)
  Interventions: Drug: nasal mupirocin; Drug: topical 3% hexachlorophene body wash; Drug: oral anti-MRSA antibiotic

INTERVENTIONS:
Drug: nasal mupirocin — twice daily for 10 days
  Other Names: Bactrban Nasal
Drug: topical 3% hexachlorophene body wash — daily for 10 days
  Other Names: Phisohex
Drug: oral anti-MRSA antibiotic — The choice of oral antibiotic was based on investigators choice and antibiotic susceptibility of prior MRSA isolates in a given patient
  Other Names: trimethoprim-sulfamethoxazole; doxycycline; minocycline

SUMMARY:
This clinical trial tests the hypothesis that body decolonization of patients with recurrent community-associated (CA) MRSA infections will significantly reduce the likelihood of recurrent CA-MRSA infection.

DETAILED DESCRIPTION:
Staphylococcus aureus is a ubiquitous pathogen, and causes infections of the skin, lung, bloodstream, and other body parts. Over the past decade,community-acquired methicillin resistant S. aureus (CA-MRSA) infections, which were previously extremely rare, are occurring commonly worldwide. CA-MRSA is the most common cause of skin infection in many locales in the U.S.

CA-MRSA strains are notable for their ability to spread in closed settings and cause recurrent infections among healthy persons. Management of recurrent CA-MRSA infection is challenging and optimal prevention strategies are undefined. Many experts recommend topical agents that decontaminate the body and/or anterior nares. However, there are no data that quantify the efficacy and safety of this approach.

We conducted a prospective non-comparative clinical trial to quantify the efficacy and safety of body decolonization regimens in the prevention of CA-MRSA infection from an Infectious Diseases private practice group in Northern California.

The study population comprised of persons suffering from recurrent CA-MRSA infection. For this clinical trial, all subjects will be given: nasal mupirocin (Bactroban Nasal, twice daily), topical 3% hexachlorophene body wash (Phisohex, daily), and an oral anti-MRSA antibiotic. The choice of oral antibiotic was based on investigators choice and antibiotic susceptibility of prior MRSA isolates in a given patient.

Patients were interviewed in person baseline and by phone at 2 weeks, 3 months, and 6 months using a standardized questionnaire. The baseline survey, based on a previously developed instrument used for an epidemiologic investigation of MRSA asked about MRSA risk factors and health-related quality of life. Follow up surveys asked about adverse drug effects, especially gastrointestinal and dermatologic side effects (2 week visit only) and incident skin and MRSA infections.

ELIGIBILITY:
Inclusion Criteria: recurrent MRSA infections and had greater than or equal to 2 MRSA infections in the 6 months prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
A new MRSA or skin infection consistent with MRSA infection. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Allen Radner, M.D., Principal Investigator — Navidad Medical Center